CLINICAL TRIAL: NCT05008042
Title: Evaluation of the Efficiacy of Mecobalamine (Vit B12) in the Treatment of Long-term Pain in Women Diagnosed With Fibromyalgia: Single-blind Randomized Controlled Trial With Three-month Follow up
Brief Title: Evaluation of the Efficiacy of Mecobalamine in the Treatment of Long-term Pain in Women Diagnosed With Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Linnaeus University (Other)
Collaborators: Landstinget i Kalmar Län (Other); Region Östergötland (Other); Karolinska Institutet (Other); Kronoberg County Council (Other Government)
Responsible Party: Principal Investigator, Carina Elmqvist, Associate professor, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRACT 2015-005086-23
Record Dates: First submitted 2021-06-30; First posted 2021-08-17 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia,; Chronic pain,; Mekobalamin,; Randomized Controlled Trial; VitaminB12
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — mecobalamin

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with Three-month follow up
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mecobalamine 5 mg/ml (Active Comparator): The active substance of vitamin B12 given in the study is Mecobalamin 5mg / ml 2 ml ie 10 mg and is given intramuscularly.
  Interventions: Drug: Mecobalamin 5 MG
- NaCl 9mg/ml (Placebo Comparator): Placebo substance given in the study is Sodium Chloride (NaCL) 9 mg / ml 2 ml, isotonic solution for parenteral use (Baxter) given intramuscularly.
  Interventions: Other: Placebo Comparator : NaCl 9 mg/ml

INTERVENTIONS:
Drug: Mecobalamin 5 MG — The Active substance of vitamin B12 is Mecobalamin 5 mg/ml is given intramuscularly
  Arms: Mecobalamine 5 mg/ml
Other: Placebo Comparator : NaCl 9 mg/ml — Sodium Chloride (NaCL) 9 mg / ml 2 ml, isotonic solution for parenteral use (Baxter) is given intramuscularly.
  Arms: NaCl 9mg/ml

SUMMARY:
Fibromyalgia causes long term pain where mostly women are affected. It is not entirely clear how vitamin B12 affects the human pain system, there are however many primary studies that indicate different interesting approaches. Considering that the receptor of NMDA is involved in both long-term pain and vitamin B12 deficiency its of most importance to evaluate whether vitamin B12 decreases the pain sensitivity and the experience of pain i.e hyperalgesia and allodynia, at persons with fibromyalgia.The aim of this study is therefore to evaluate the effect of Mecobalamin (vitamin B12), and describe lived experiences of pain, health, suffering and well-being in women with diagnosed fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-70 years
* Swedish-speaking
* Diagnosis of fibromyalgia
* Safe method of contraception
* Cobalamin / p (vitamin B12) should be >250 pmol/L < 800 pmol/L
* Given consent to participate.

Exclusion Criteria:

* Previous treatment with B12
* Known hypersensitivity to the active substance Mecobalamin or an additive
* Vegan as veganism can lead to B12 deficiency
* Neuroleptics
* Known heart, kidney or liver disease
* Reynaud's phenomenon (white fingers)
* Known neuropathy (impaired sensation)
* Breastfeeding
* Pregnancy or plan pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Tolerance time | 24 weeks
  Primary outcome is tolerance time, maximized to Three minutes, tested using the Cold Pressure test

SECONDARY OUTCOMES:
Pain experience measured by a pressure algometry test | 24 weeks
  Pain experience measured by a pressure algometry test performed on the shoulder, hip, knee and elbow.
Possible pain change measured by a pressure algometry test | 24 weeks
  Possible pain change measured by a pressure algometry test performed on the shoulder, hip, knee and elbow.
Subjective experience of pain measured using Numeric Rating Scale (NRS) | 24 weeks
  Subjective experience of pain measured using Numeric Rating Scale (NRS) 0-10 where 0 is the best outcome .
Possible pain change measured using Numeric Rating Scale (NRS) 0-10 | 24 weeks
  Possible pain change measured using Numeric Rating Scale (NRS) 0-10 where 0 is the best outcome .
Ratings of expectation, desire for relief, using Numeric Rating Scale (NRS) | 24 weeks
  Ratings of expectation, desire for relief, using Numeric Rating Scale (NRS) 0-10 where 0 is the best outcome.
Ratings of expectation, pain variability, using Numeric Rating Scale (NRS) 0-10 | 24 weeks
  Ratings of expectation, pain variability, using Numeric Rating Scale (NRS) 0-10 where 0 is the best outcome.
Activity level, assessed using questionnaire McGills Pain Questionnaire (MPQ). | 24 weeks
  Activity level are assessed using questionnaire McGills Pain Questionnarie (MPQ). Short version score 0-45.
Quality of Life are assessed using questionnaires RAND-36. | 24 weeks
  Quality of life are assessed using questionnaires RAND-36 score 0-100
Experience of the effect of the drug, assessed using questionnaire Patients´ Global Impression of Change (PGIC). | 24 weeks
  Experience of the effect of the drug, score 1-7
Cobalamin in plasma | 24 weeks
  Control of vitamin B12 is done by measuring cobalamin in plasma.
Lived experiences of pain, health, suffering and well-being. | 24 weeks
  Qualitative in-depth interviews will be conducted to capture women's lived experiences of pain, health, suffering and well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Carina Elmqvist, Ass prof, Principal Investigator — Linnaeus University
Locations (1):
- Linnaeus University, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Metadata and analysis scripts
Supporting Information: Study Protocol, SAP, ICF
Time Frame: from 2025 - 2035
Access Criteria: anyone requesting the metadata can access the data

REFERENCES:
- [Derived] Sall Hansson K, Lindqvist G, Stening K, Fohlman J, Wojanowski A, Ponten M, Jensen K, Gerdle B, Elmqvist C. Efficacy of mecobalamin (vitamin B12) in the treatment of long-term pain in women diagnosed with fibromyalgia: protocol for a randomised, placebo-controlled trial. BMJ Open. 2023 Mar 30;13(3):e066987. doi: 10.1136/bmjopen-2022-066987. PMID 36997252